CLINICAL TRIAL: NCT01841242
Title: Comparison of Alcoholic Chlorhexidine 2% Versus Alcoholic Povidone Iodine for Infections Prevention With Cardiac Resynchronization Therapy Device Implantation
Acronym: CHLOVIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government); C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1108096; 2012-000803-33 (EudraCT Number)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Arrhythmia
Keywords: Infection; Cardiac Resynchronization Device; Heart Failure
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Infections

STUDY DESIGN:
Intervention Model Description: 2 randomized groups
Oversight: Data Monitoring Committee: No

ARMS (2):
- alcoholic povidone iodine (Active Comparator): Betadine Alcoolique 5% One cutaneous application before implant procedure
  Interventions: Drug: alcoholic povidone iodine
- alcoholic chlorhexidine (Experimental): ChloraPrep 2% One cutaneous application before implant procedure
  Interventions: Drug: alcoholic chlorhexidine

INTERVENTIONS:
Drug: alcoholic povidone iodine
  Other Names: Betadine alcoolique 5%
  Arms: alcoholic povidone iodine
Drug: alcoholic chlorhexidine
  Other Names: ChloraPrep 2%
  Arms: alcoholic chlorhexidine

SUMMARY:
Heart Failure (HF) with systolic dysfunction is associated with a poor prognosis in the long term despite the use of many effective drug treatment in reducing morbidity and mortality. In this context, cardiac resynchronization (CR), either alone or combined with a defibrillator function, has improved by about 30 to 40% of morbidity and mortality in this population of patients with heart failure. The information on the CR are now well established for patients with stage III-IV NYHA (New York Heart Association), with systolic dysfunction (EF ≤ 35%), presence of left bundle branch block wide (≥ 120 ms) and when medical treatment is optimal. As a result, the number of implanted devices continue to grow even if the implant procedures of cardiac resynchronization devices (CRD) are long, difficult and associated with significant complications with a risk of reoperation estimated between 10 and 15% . One of the most feared during implantation devices stimulation or defibrillation risk is represented by the risk of infection that will lead inevitably to explantation of the device. Despite the use of several preventive measures, including the use of an antiseptic shower, a local preparation for alcoholic povidone iodine (API) (PVPI 5% ethanol + 70%) and antibiotic prophylaxis clinical studies the most recent have clearly demonstrated that the risk of infection was associated with the duration of the intervention and was higher for procedures CR, it is noted in 2.4% in the short term and would be close to 3 to 4% in the medium term. Infections of implantable devices are associated with a poor prognosis, even in an excess mortality. It has been shown that the majority of infections may be linked to local contamination during surgery reinforcing the idea that prevention is mainly based on local measures and the reduction of operating time.

DETAILED DESCRIPTION:
In this context, all measures that will reduce the risk of infection, will improve the prognosis of these patients. Thus, recent studies have shown greater effectiveness of local preparation for alcoholic chlorhexidine (applicator containing 2% chlorhexidine and 70% alcohol isopropanolol) (AC 2%) compared to the aqueous povidone iodine (API)in general surgery. It has been shown that the rate of local infection was significantly reduced in the AC group vs 2%. aqueous povidone iodine, respectively vs. 9.5%. 16.1% (p = 0.004). No randomized trials have previously prospectively compared the interest of local preparation with AC 2% compared with the usual preparation by API during implantation Resynchronization devices. Based on experimental and clinical studies, and we hope this new approach to assess local skin preparation in the prevention of general and local risk of infection after implantation of a cardiac resynchronization device. To ensure consistency, and because of its high efficiency assumed on the basis of experimental and clinical studies, the choice fell on the revenue 2% with applicator and patients should benefit from a primary location or "up-grading" to a CR device.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring cardiac resynchronization therapy (stage III-IV NYHA, EF ≤ 35%, left bundle branch block large (≥ 120 ms), optimal medical therapy) OR patients requiring the implementation of a resynchronization device on basis of the study PAVE (FE ≤ 45% + Atrial Fibrillation + need a radiofrequency atrioventricular node) OR patients requiring implantable pacemaker or implantable defibrillator but NYHA stage II, EF ≤ 35%; branch block left large (≥ 150 ms) optimal medical treatment OR patient requiring an upgrading at least 2 years after their last implementation
* Patient has consented free, informed
* Patients whose prognosis is not compromised by a morbid pathology in one year
* absence of contraindication to povidone-iodine alcoholic
* absence of contraindication to 2% chlorhexidine in alcohol or yellow-orange S (E110)

Exclusion Criteria:

* Change case of cardiac resynchronization
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2272 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Infection | 24 months
  Local or general infection in relation to the implantable device (skin erosion, externalization, local flow, local abscess, sepsis with or without bacteremia)

SECONDARY OUTCOMES:
Cardiovascular event | 24 months
  Major cardiovascular events such as heart failure, embolic right heart.
Side Effects | 24 months
  Side effects attributable to local treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DA COSTA, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (24):
- France (24):
  - CH d'Aix en Provence, Aix-en-Provence
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d'Annecy, Annecy
  - CH d'Avignon, Avignon
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CH de Chartres, Chartres
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CH la Rochelle, La Rochelle
  - CHU de Lille, Lille
  - Ch St Joseph St Luc, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - CH de Périgueux, Périgueux
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Da Costa A, Mansourati J, Eschalier R, Lesaffre F, Bordachar P, Taieb J, Laurent G, Milhem A, Kubala M, Le Page S, Milliez P, Gal B, Dompnier A, Defaye P, Bayle S, Anselme F, Cheggour S, Litalien J, Duparc A, Pasquier JL, Romeyer C, Botelho-Nevers E, Gagnaire J, Lager E, Garcin A, Chapelle C, Schimd A, Benali K, Laporte S, Deharo JC; CHLOVIS Study Investigators. Chlorhexidine vs Povidone-Iodine Alcohol Solutions for Cardiac Implantable Electronic Devices: A Prospective Randomized Study. J Am Coll Cardiol. 2026 Jan 20;87(2):200-211. doi: 10.1016/j.jacc.2025.10.042. PMID 41562534